CLINICAL TRIAL: NCT03281655
Title: Effects of a New Vaginal Cream Containing Visnadine, Prenylflavonoids and Bovine Colostrum in Postmenopausal Sexually Active Women Affected by Vulvovaginal Atrophy: a Prospective Cohort Analysis
Brief Title: Visnadine, Prenylflavonoids and Bovine Colostrum to Treat Vulvovaginal Atrophy in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Messina (Other)
Collaborators: University of Victoria (Other); University of Athens (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REFEEL-1
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Vulvovaginal Atrophy; Menopause
Keywords: Visnadine; Prenylflavonoids; Bovine colostrum; Sexual wellbeing
MeSH Terms: interventions — visnadin

STUDY DESIGN:
Intervention Model Description: Single cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vulvovaginal atrophy (Experimental): Postmenopausal sexually active women affected by vulvovaginal atrophy undergoing treatment (15 days, 1 application per day) with a vaginal cream containing visnadine, prenylflavonoids and bovine colostrum.
  Interventions: Drug: Visnadine, prenylflavonoids and bovine colostrum

INTERVENTIONS:
Drug: Visnadine, prenylflavonoids and bovine colostrum — 15 days, 1 application per day, with a vaginal cream containing visnadine, prenylflavonoids and bovine colostrum.

SUMMARY:
The effects of a new vaginal cream containing visnadine (0.30%), prenylflavonoids (0.10%) and bovine colostrum (1%) will be evaluated in post-menopausal sexually active women affected by vulvovaginal atrophy (VVA).

In a prospective cohort study, post-menopausal women affected by VVA will be enrolled. All women will undergo vaginal health index score (VHIS) evaluation and will complete the female sexual function index (FSFI) questionnaire at baseline evaluation (T0) and following 15 days of vaginal cream treatment with one application per day (T1). All the side effects will be recorded and an independent data safety and monitoring committee will evaluate the results of the study.

DETAILED DESCRIPTION:
Sexual health plays a key role during women's lives from puberty to post-menopausal period and, for this reason, it has increasingly received public health, pharmaceutical, and medical attention. According to the study of women's health across the nation (SWAN), more than 75% of the middle-aged women reported that sex was moderately to extremely important; in addition, the menopausal transition was characterized by increasing pain during sexual intercourse and consequent decrease of sexual desire. Individual general health status, diabetes mellitus, cardiovascular diseases, other genitourinary diseases, psychiatric/psychological disorders, other chronic diseases and socio-demographic conditions may all influence post-menopausal sexual health. Although aging could be considered an independent risk factor for sexual dysfunction accumulating evidence suggests that vulvovaginal atrophy (VVA) is strongly associated with female sexual dysfunction (FSD) among sexually active postmenopausal women: in particular, VVA was found to be significantly associated with a global indication of FSD and difficulties with sexual desire, arousal, and orgasm. VVA often results from postmenopausal estrogen loss, which acts as a double-edged sword: on the one hand, it plays a detrimental action on woman's desire and arousal; on the other hand, it decreases the lubrication of the vagina before sexual activity and, consequently, causes pain during intercourse, precludes satisfaction and further decreases arousal.

Although several pharmacological approaches have been evaluated for the relief of VVA. Local estrogens are considered a safe option for VVA, although many clinicians are hesitant to prescribe them and many women reluctant to use them. In addition, non-hormonal treatments such as moisturizers and precoital vaginal lubricants could be considered a safer alternative, even in cancer patients. In this regard, visnadine, an active ingredient of the fruit of Ammi visnaga, showed powerful vasodilatory activity, due to the inhibitory effects on vascular smooth muscles mediated by Ca2+ entry through voltage-gated L-type Ca2+ channels. In addition, visnadine improves both female sexual function index (FSFI) and color Doppler sonography of clitoral blood flow. Furthermore, prenylflavonoids and phytoestrogens play a potent role as estrogen receptor (ER)-alpha selective agonist, thus they may counteract the effects of postmenopausal estrogen loss. Finally, a vaginal cream containing bovine colostrum has been shown to be effective in relieving vaginal dryness and other VVA symptoms in postmenopausal women, after 8 weeks of treatment. Based on this information, the investigators aim to evaluate the effects of a new vaginal cream containing visnadine, prenylflavonoids and bovine colostrum on vaginal health index score (VHIS) and FSFI in a cohort of postmenopausal sexually active women affected by VVA.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal sexually active women affected by vulvovaginal atrophy.

Exclusion Criteria:

* relevant comorbidities (chronic cardiovascular, immune, endocrine and metabolic diseases and cancers);
* smokers;
* who used any other kind of pharmacologic treatment (including the substances tested in this study) in the previous 3 months.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Vaginal health index score (VHIS) evaluation | Post-treatment (15 days)
  Elasticity, fluid volume and consistency, pH, epithelial integrity and moisture.
Female sexual function index (FSFI) questionnaire | Post-treatment (15 days)
  Desire, arousal, lubrication, orgasm, satisfaction and pain.

SECONDARY OUTCOMES:
Side effects | Post-treatment (15 days)
  Number of side effects during/after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — University of Messina; Salvatore Giovanni Vitale, M.D., Principal Investigator — University of Messina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slater C, Robinson AJ. Sexual health in adolescents. Clin Dermatol. 2014 Mar-Apr;32(2):189-95. doi: 10.1016/j.clindermatol.2013.08.002. PMID 24559553
- [Background] Schwenkhagen A. Hormonal changes in menopause and implications on sexual health. J Sex Med. 2007 Mar;4 Suppl 3:220-6. doi: 10.1111/j.1743-6109.2007.00448.x. PMID 17394594
- [Background] McCabe MP, Sharlip ID, Lewis R, Atalla E, Balon R, Fisher AD, Laumann E, Lee SW, Segraves RT. Incidence and Prevalence of Sexual Dysfunction in Women and Men: A Consensus Statement from the Fourth International Consultation on Sexual Medicine 2015. J Sex Med. 2016 Feb;13(2):144-52. doi: 10.1016/j.jsxm.2015.12.034. PMID 26953829
- [Background] Avis NE, Brockwell S, Randolph JF Jr, Shen S, Cain VS, Ory M, Greendale GA. Longitudinal changes in sexual functioning as women transition through menopause: results from the Study of Women's Health Across the Nation. Menopause. 2009 May-Jun;16(3):442-52. doi: 10.1097/gme.0b013e3181948dd0. PMID 19212271
- [Background] Avis NE, Colvin A, Bromberger JT, Hess R, Matthews KA, Ory M, Schocken M. Change in health-related quality of life over the menopausal transition in a multiethnic cohort of middle-aged women: Study of Women's Health Across the Nation. Menopause. 2009 Sep-Oct;16(5):860-9. doi: 10.1097/gme.0b013e3181a3cdaf. PMID 19436224
- [Background] Dennerstein L, Hayes RD. Confronting the challenges: epidemiological study of female sexual dysfunction and the menopause. J Sex Med. 2005 Sep;2 Suppl 3:118-32. doi: 10.1111/j.1743-6109.2005.00128.x. PMID 16422789
- [Background] Hayes R, Dennerstein L. The impact of aging on sexual function and sexual dysfunction in women: a review of population-based studies. J Sex Med. 2005 May;2(3):317-30. doi: 10.1111/j.1743-6109.2005.20356.x. PMID 16422862
- [Background] Levine KB, Williams RE, Hartmann KE. Vulvovaginal atrophy is strongly associated with female sexual dysfunction among sexually active postmenopausal women. Menopause. 2008 Jul-Aug;15(4 Pt 1):661-6. doi: 10.1097/gme.0b013e31815a5168. PMID 18698279
- [Background] Nappi RE, Palacios S, Particco M, Panay N. The REVIVE (REal Women's VIews of Treatment Options for Menopausal Vaginal ChangEs) survey in Europe: Country-specific comparisons of postmenopausal women's perceptions, experiences and needs. Maturitas. 2016 Sep;91:81-90. doi: 10.1016/j.maturitas.2016.06.010. Epub 2016 Jun 15. PMID 27451325
- [Background] Castelo-Branco C, Biglia N, Nappi RE, Schwenkhagen A, Palacios S. Characteristics of post-menopausal women with genitourinary syndrome of menopause: Implications for vulvovaginal atrophy diagnosis and treatment selection. Maturitas. 2015 Aug;81(4):462-9. doi: 10.1016/j.maturitas.2015.05.007. Epub 2015 May 30. PMID 26071816
- [Background] Lethaby A, Ayeleke RO, Roberts H. Local oestrogen for vaginal atrophy in postmenopausal women. Cochrane Database Syst Rev. 2016 Aug 31;2016(8):CD001500. doi: 10.1002/14651858.CD001500.pub3. PMID 27577677
- [Background] Derzko C, Elliott S, Lam W. Management of sexual dysfunction in postmenopausal breast cancer patients taking adjuvant aromatase inhibitor therapy. Curr Oncol. 2007 Dec;14 Suppl 1(Suppl 1):S20-40. doi: 10.3747/co.2007.151. PMID 18087605
- [Background] Bassino E, Antoniotti S, Gasparri F, Munaron L. Effects of flavonoid derivatives on human microvascular endothelial cells. Nat Prod Res. 2016 Dec;30(24):2831-2834. doi: 10.1080/14786419.2016.1154053. Epub 2016 Mar 2. PMID 26936689
- [Background] Caruso S, Mauro D, Cariola M, Fava V, Rapisarda AMC, Cianci A. Randomized crossover study investigating daily versus on-demand vulvar Visnadine spray in women affected by female sexual arousal disorder. Gynecol Endocrinol. 2018 Feb;34(2):110-114. doi: 10.1080/09513590.2017.1354366. Epub 2017 Jul 27. PMID 28749253
- [Background] Schaefer O, Humpel M, Fritzemeier KH, Bohlmann R, Schleuning WD. 8-Prenyl naringenin is a potent ERalpha selective phytoestrogen present in hops and beer. J Steroid Biochem Mol Biol. 2003 Feb;84(2-3):359-60. doi: 10.1016/s0960-0760(03)00050-5. No abstract available. PMID 12711023
- [Background] Nappi RE, Cagnacci A, Becorpi AM, Nappi C, Paoletti AM, Busacca M, Martella S, Bellafronte M, Tredici Z, Di Carlo C, Corda V, Vignali M, Bagolan M, Sardina M. Monurelle Biogel(R) vaginal gel in the treatment of vaginal dryness in postmenopausal women. Climacteric. 2017 Oct;20(5):467-475. doi: 10.1080/13697137.2017.1335703. Epub 2017 Jun 28. PMID 28657769